CLINICAL TRIAL: NCT07182305
Title: Treatment Trial With Albendazole of Patients With a Diagnosis of Early Stage Alveolar Echinococcosis
Brief Title: Treatment Trial of Alveolar Echinococcosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ministry of Health, Kyrgyzstan (Other Government)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Gulnara Minbaeva, Epidemiologist, Ministry of Health, Kyrgyzstan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AE-Kyrgyzstan
Record Dates: First submitted 2017-05-22; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Alveolar Echinococcosis
Keywords: alveolar echinococcosis; Echinococcus multilocularis; albendazole
MeSH Terms: conditions — Alveolar echinococcosis; Echinococcosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Cases defined as early stage alveolar echinococcosis receive daily dose of albendazole 2 x 400 mg
  Interventions: Drug: Efficacy of albendazole for early stage intervention of alveolar echinococcosis
- Control (No Intervention): Cases defined as early stage alveolar echinococcosis not receiving placebo treatment

INTERVENTIONS:
Drug: Efficacy of albendazole for early stage intervention of alveolar echinococcosis — Participants in the treatment arm will be treated with albendazole, 2 x 400 mg daily for the duration of the study. Treatment may be prolonged beyond the end of the study if clinically appropriate.
  Arms: Treatment

SUMMARY:
A new focus of subjects with lesions of alveolar echinococcosis caused by Echinococcus multilocularis has been found south of Gulcha in Osh province in Kyrgyzstan by an ultrasound surveillance. Prevalence of infections is approximately 6%. Most lesions are small. Current scientific evidence suggests that in the absence of treatment, alveolar echinococcosis has a case fatality rate approaching 100% within 10-15 years of infection. Albendazole is known to be effective as a parasitostatic treatment to prolong the life of subjects with this disease, possibly up to normal life expectancy with prolonged treatment. The trial will be a case control study to evaluate the treatment of subjects with early stage alveolar echinococcosis and the progression of disease.

DETAILED DESCRIPTION:
1. case definition of patients with early stage alveolar echinococcosis. These are patients who are otherwise healthy, but have been identified as having hepatic lesions consistent with alveolar echinococcosis as diagnosed by ultrasound through a monitoring programme.
2. Subjects will be randomised 60 patients into treatment and 60 into non treatment groups.
3. Randomisation should be such that approximately similar age and gender profiles match in each group.
4. Baseline examination by imaging. Define the lesion and case definition. Blood samples taken from all subjects at baseline
5. Blood is analysed for serological evidence of echinococcosis
6. Treatment is started. Treatment for case group is 2 x 400 mg Albendazole, daily. Control group has a placebo.
7. Monitor at 2 weeks and 4 weeks for liver function, serology and imaging
8. Monitor every 3 months thereafter.
9. Subjects that have any evidence of lesion progression will be referred for surgical treatment regardless of treatment group.
10. Monitoring for 2 years. Assess lesions in treatment and placebo groups. Assess dynamics of antibody (if any). Assess numbers of subjects from each group who have been referred for surgery following progression of lesion.
11. Indicators for premature ending of trail would include evidence that the treatment is effective (ie treatment group not progressing or lesions regressing, whilst non treatment group lesions increase in size) - action all subjects now put into therapy.

No effect of albendazole - lesions progressing in all cases - indicating surgical treatment required in all cases.

Most lesions regressing in both the treatment and control group - indicates most early cases spontaneously resolve. Stop treatment but continue to monitor all cases.

ELIGIBILITY:
Inclusion Criteria:

* Presence of lesion diagnosed by ultrasound that is consistent with early stage alveolar echinococcosis. Lesion less than 3 cm in diameter

Exclusion Criteria:

* Absence of lesion. Large lesion requiring surgical treatment

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Progression of parasitic lesion | 3 years
  Increase in size of lesion or regression or calcification. Participants will be regularly assessed using ultrasound imaging of the lesion. The lesion size will me measured. The size of the lesion was measured using the cross-sectional image with the longest diameter on ultrasound. The measurement will be in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Gulnara Minbaeva, MD, Principal Investigator — Department of disease prevention and sanitary - epidemiological surveillance, Ministry of Health of the Kyrgyz Republic
Locations (1):
- Department of disease prevention and sanitary - epidemiological surveillance, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: No
IPD will be confidential or anonymised. Results will be published but no patient will be identifiable. Such will be freely available from mid 2019 and available between the trial investigators from the start of the trial